CLINICAL TRIAL: NCT05232175
Title: A Phase I Study to Evaluate the Tolerance, Safety and Pharmacokinetics of ALT-BB4 in Healthy Volunteer
Brief Title: Clinical Study of ALT-BB4 to Determine Tolerance, Safety and Pharmacokinetics in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alteogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-BB4-01
Record Dates: First submitted 2022-01-14; First posted 2022-02-09 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Health, Subjective
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part I (Allergy assessment) - ALT-BB4 (Experimental)
  Interventions: Drug: ALT-BB4
- Part I (Allergy assessment) - 0.9%NaCl (Placebo Comparator)
  Interventions: Drug: 0.9%NaCl
- Part II-A (PK assessment) (Experimental)
  Interventions: Drug: ALT-BB4
- Part II-B (Safety assessment) - ALT-BB4 (Experimental)
  Interventions: Drug: ALT-BB4
- Part II-B (Safety assessment) - 0.9% NaCl (Placebo Comparator)
  Interventions: Drug: 0.9%NaCl

INTERVENTIONS:
Drug: ALT-BB4 — Recombinant Hyaluronidase
  Arms: Part I (Allergy assessment) - ALT-BB4; Part II-A (PK assessment); Part II-B (Safety assessment) - ALT-BB4
Drug: 0.9%NaCl — Normal Saline
  Arms: Part I (Allergy assessment) - 0.9%NaCl; Part II-B (Safety assessment) - 0.9% NaCl

SUMMARY:
A Phase I Study to Evaluate the Tolerance, Safety and Pharmacokinetics of ALT-BB4 in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

Common

1. Healthy volunteers aged ≥19 years at the time of Screening (Visit 1)
2. Female subjects or male subjects' female partner must be menopausal or should have received a sterilization procedure or have agreed to use contraceptive methods during the study period, as defined below:

   * Post-menopausal female subjects or male subjects' female partners (non-drug induced amenorrhea for at least 12 months or confirmed diagnosis with menopause)
   * Female subjects or male subjects' female partners who have received a sterilization procedure (removal of ovary and/or uterus)
   * Subjects who have agreed to practice total abstinence during the study period [For female subjects, periodic abstinence (e.g., ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.]
   * When female subjects or male subjects' female partners are women of childbearing potential (WOCBP) who have not received a sterilization procedure, they must agree to use of following contraceptive methods:
   * Hormones (implantable, patch, and oral)
   * Intrauterine device (IUD)
   * Double barrier methods (concomitant use of two of following contraceptive methods: male condom, female condom, cervical cap, diaphragm, sponge, spermicide) (However, concomitant use of male condom and female condom is excluded from double barrier methods.)
3. WOCBP or females who have the last menstrual period within 12 months must have a negative serum or urine pregnancy test at Screening (Visit 1).
4. Subjects who have voluntarily decided to take part in the study and able to comply with the study protocol
5. Subjects who have no tattoo, acne, dermatitis, pigmentation or lesion on the administration site and who have no damage in the skin, so that they can receive the IP and allergy test
6. Subjects determined eligible for the study through Screening tests (vital signs, physical examination, medical history and surgery history, ECG, and laboratory tests)

   Part II-A
7. Subjects with BMI no less than 18.5 kg/m2, no greater than 24.9 kg/m2

Exclusion Criteria:

Common

1. Subjects who have received or treated with following medications within the specified timeframe prior to Screening (Visit 1) or who are expected to receive them during the study period:

   * Within 1 month: Hyaluronidase, Chemotherapeutic agent, non-steroidal anti-inflammatory drugs (NSAIDs; e.g.: Aspirin, Aceclofenac, etc.), penicillins antibiotics (e.g.: Amoxicillin, Ampicillin, etc.), cephalosporins antibiotics (e.g.: Cefaclor, Cefadroxil, Cefixime, etc.), sulfonamides antibiotics (e.g.: Sulfadiazine, Sulfamethoxazole, etc.), quinolones antibiotics (e.g.: Ciprofloxacin, Levofloxacin, etc.), Glucocorticosteroid, Immunosuppressive agent
   * Within 14 days: Antihistamine (e.g.: Chlorpheniramine, Hydroxyzine, Ketotifen, etc.)
2. Subjects who have prior history of clinically significant liver, kidney, nervous system, immune system, respiratory system, endocrine system, hematology/neoplasm, cardiovascular system, mental (mood disorder, obsessive-compulsive disorder), gastrointestinal disorders or surgical history
3. Subjects with acute fever > 37.5℃ within 7 days from the expected IP administration or showing symptoms suspecting acute diseases within 14 days from the expected IP administration
4. Subjects who do not have normal blood pressure*

   *Range of normal blood pressure is defined as systolic and diastolic blood <120/80 mmHg in accordance with 2018 Korean Society of Hypertension Guidelines for the Management of Hypertension24) (however, Pre-hypertension (≥ 130/80) is excluded that may occur in normotension).
5. Subjects who persistently drink more than the weekly recommended alcohol units* 14 g of alcohol content per unit is applied, which corresponds to 1 can (small bottle) of beer (5%), 350 mL of draft beer (5%), 1 cup (300 mL) of makgeoli, 1 glass (150 mL) of wine (12%), 1/4 bottle (90 mL) of soju (20%), and 1 shot (45 mL) of liquor (40%). Moderate amount of alcohol by age and gender is provided below:23) Age Recommended unit per week Adults (≥ 19 and < 65 years) Male: 8 units/week Female: 4 units/week Elderly (≥ 65 years) Male: 4 units/week Female: 2 units/week
6. Subjects of usual smoker (exceeding 10 cigarettes per day)
7. Subjects who have a past history of autoimmune diseases (e.g.: rheumatoid arthritis, etc.) or active immune diseases that may affect the immune system [e.g.: flu, cancer, Human immunodeficiency virus (HIV), Hepatitis B virus (HBV), Hepatitis C virus (HCV) etc.], diabetes mellitus, heart diseases, asthma, sinusitis, chronic urticaria, dermographism, or any skin conditions that may affect post-IP administration assessments (e.g.: Dermatitis, dermatomycosis and other skin diseases or tattoo)
8. Subjects with known allergic reactions or hypersensitivity to bee sting or other common allergens or known contraindications to hyaluronidase, thimerosal (disinfectants) and EDTA
9. Subjects with hypersensitivity to the IP or its ingredients or a history of anaphylaxis
10. Past history of drug abuse
11. Subjects who have participated in other clinical trials within 6 months prior to the expected IP administration
12. Others determined ineligible for the study participation in the opinion of investigator

    Part II-A
13. Subjects who have been treated with a drug-metabolizing enzyme inducers and inhibitors*25), 26) within 30 days prior to the IP administration

    * Example: Phenytoin, Carbamazepine, Barbiturates, Rifampicin, Griseofulvin, Cimetidine, Disulfiram, Erythromycin, Ketoconazole, Fluconazole, Itraconazole, Valproic acid, Isoniazid, Ciprofloxacin, Omeprazole, Clarithromycin, Quinidine, Sulfonamides, etc.
14. Subjects who have significant bleeding or blood loss within 60 days prior to Screening (Visit 1)
15. Subjects who have donated whole blood within 60 days or donated blood by apheresis within 14 days or received transfusion within 14 days prior to Screening (Visit 1)
16. Subjects who have consumed grapefruit juice28) within 7 days prior to Screening (Visit 1)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Derived] Lee JS, Kim W, Won CH, Lee YW, Lee S, Won H, Park SJ, Lee S, Kim SH, Yang J, Bahn G, Lee DH. The Safety, Tolerability, and Pharmacokinetics of ALT-BB4 (A Novel Recombinant Hyaluronidase): A Randomized, Double-Blinded, Placebo-Controlled, Phase 1 Study in Healthy Volunteers. Dermatol Ther (Heidelb). 2025 Nov;15(11):3301-3311. doi: 10.1007/s13555-025-01507-x. Epub 2025 Sep 2. PMID 40892310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in four sites in the Republic of Korea from January 18, 2022, to August 24, 2022.
Pre-assignment Details: The study consisted of Part I and Part Ⅱ, and a total of 244 participants received study treatments. Among the 290 enrolled participants, 46 were excluded from the Part 1 safety analysis due to an injection-site randomization error.
Units Other Than Participants: Forearms
Groups:
- All Study Participants: PartⅠ(Allergy assessment): Participants were randomly assigned to receive intradermal administrations of ALT-BB4 or placebo into either the right or left forearm.
  Part Ⅱ-A (PK assessment): Participants in Part Ⅱ-A included only subjects who had a negative drug allergy in the PartⅠ.
  ALT-BB4 was administered subcutaneously into either the left or right upper arm.
  PartⅡ-B (Safety assessment): Participants in Part Ⅱ-B included only subjects who had a negative drug allergy in the PartⅠ.
  Enrolled subjects were randomized in a 2:1 ratio to receive ALT-BB4 or the comparator.
  Investigator products (IP) were administered subcutaneously into either the right or left upper arm.
Period: Part I (Allergy assessment)
Arm/Group | All Study Participants
Started | 244; 488 Forearms
ALT-BB4 | 244; 244 Forearms
Placebo | 244; 244 Forearms
Completed | 244; 488 Forearms (Seven participants were discontinued from the study after completing Part I and did not proceed to Part II)
Not Completed | 0; 0 Forearms
Period: Part Ⅱ-A (PK assessment)
Arm/Group | All Study Participants
Started | 23; 23 Forearms
Completed | 23; 23 Forearms
Not Completed | 0; 0 Forearms
Period: PartⅡ-B (Safety assessment)
Arm/Group | All Study Participants
Started | 214; 214 Forearms
ALT-BB4 | 142; 142 Forearms
Placebo | 72; 72 Forearms
Completed | 214; 214 Forearms
Not Completed | 0; 0 Forearms

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomly assigned to receive intradermal administrations of ALT-BB4 or placebo into either the right or left forearm.
  Participants in Part Ⅱ-A included only subjects who had a negative drug allergy in the PartⅠ.
  ALT-BB4 was administered subcutaneously into either the left or right upper arm.
  Participants in Part Ⅱ-B included only subjects who had a negative drug allergy in the PartⅠ.
  Enrolled subjects were randomized in a 2:1 ratio to receive ALT-BB4 or the comparator.
  Investigator products (IP) were administered subcutaneously into either the right or left upper arm.
Arm/Group | All Study Participants
Number analyzed (Participants) | 244
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 96
BMI [Mean (Standard Deviation); unit: (Kg/m2)] | 23.5 (3.6)
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 34.3 (10)
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 244

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Drug Allergy Following ID Injection of the IP
Description: Subject developing either immediate or delayed allergic reaction are considered to have drug allergy.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Groups:
- ALT-BB4; Placebo: Participants were randomly assigned to receive intradermal administrations of ALT-BB4 or placebo into either the right or left forearm.
Arm/Group | ALT-BB4 | Placebo
Number analyzed (Participants) | 244 | 244
Participants
  Immediate Drug Allergy Reaction (occurred within 30 minutes) | 0 | 0
  Delayed Drug Allergy Reaction (occurred within 48 hours) | 1 | 0

2. Primary Outcome: Injection-site TEAEs (Treatment Emergent Adverse Events)
Description: Incident rate of administration site-related adverse events in Part Ⅱ-B
Time Frame: 4 weeks
Population: In PartⅡ-B, injection site TEAEs were monitored only in subjects who tested negative for drug allergies in Part Ⅰ.
Measure: Number; unit: events
Groups:
- ALT-BB4; Placebo: Participants in Part Ⅱ-B included only subjects who had a negative drug allergy in the PartⅠ.
  Enrolled subjects were randomized in a 2:1 ratio to receive ALT-BB4 or the comparator.
  Investigator products (IP) were administered subcutaneously into either the right or left upper arm.
Arm/Group | ALT-BB4 | Placebo
Number analyzed (Participants) | 142 | 72
events | 24 | 0

ADVERSE EVENTS:
Time Frame: up to 28 days
Groups:
- PartⅠ_ALT-BB4: PartⅠ(Allergy assessment): ALT-BB4 was administered intradermally into the right or left forearm.
- PartⅠ_Placebo: PartⅠ(Allergy assessment): Placebo was administered intradermally into the right or left forearm.
- PartⅡ-A: PartⅡ-A (PK assessment): ALT-BB4 was administered subcutaneously into the left or right upper arm.
- PartⅡ-B_ALT-BB4: PartⅡ-B (Safety assessment): ALT-BB4 was administered subcutaneously into the right or left upper arm.
- PartⅡ-B_Placebo: PartⅡ-B (Safety assessment): Placebo was administered subcutaneously into the right or left upper arm.
Arm/Group | PartⅠ_ALT-BB4 | PartⅠ_Placebo | PartⅡ-A | PartⅡ-B_ALT-BB4 | PartⅡ-B_Placebo
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/244 | 0/23 | 0/142 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/244 | 0/23 | 0/142 | 0/72
Other Adverse Events (participants affected / at risk) | 61/244 | 3/244 | 6/23 | 24/142 | 0/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PartⅠ_ALT-BB4 (N=244) | PartⅠ_Placebo (N=244) | PartⅡ-A (N=23) | PartⅡ-B_ALT-BB4 (N=142) | PartⅡ-B_Placebo (N=72)
Injection site erythema (General disorders) | 51 | 2 | 3 | 17 | 0
Injection site telangiectasia (General disorders) | 8 | 0 | 0 | 6 | 0
Administration site bruise (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site urticaria (General disorders) | 1 | 1 | 0 | 1 | 0 — Injection site urticaria of ALT-BB4 group is Preferred Term, which means wheal according to MedDRA.
Injection site discolouration (General disorders) | 1 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT05232175/Prot_SAP_000.pdf